CLINICAL TRIAL: NCT02629237
Title: Impact of Multifaceted Education on Satisfaction After Glaucoma Surgery in Rural China
Brief Title: Satisfaction After Glaucoma Surgery in Rural China
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study sites were reconsidered.
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Congdon Nathan, vice directior,Blindness Prevention and Treatment Department, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ZOC-CREST-Satisfaction
Record Dates: First submitted 2015-10-09; First posted 2015-12-14 (Estimated); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Glaucoma
Keywords: glaucoma surgery; educational intervention; satisfaction; rural
MeSH Terms: conditions — Glaucoma; Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multifaceted education group (Experimental): Subjects will be asked to watch a 5-10 min education film and participate in a 10-15 min counseling session with a trained doctor/nurse before glaucoma surgery,and at 1 week and 2 week after surgery.
  Interventions: Other: Multifaceted education
- control group (No Intervention): Subjects will not be asked to watch education film and not participate in counseling session before and after surgery.

INTERVENTIONS:
Other: Multifaceted education — Subjects will be asked to watch a 5-10 min education film and participate in a 10-15 min counseling session with a trained doctor/nurse before glaucoma surgery,and at 1 week and 2 week after surgery.
  Arms: Multifaceted education group

SUMMARY:
1. Investigate degree of postoperative satisfaction in county level hospital glaucoma patients.
2. Investigate the effect of educational intervention affect the degree of satisfaction in glaucoma patients.
3. Investigate the effect factors of postoperative satisfaction.

DETAILED DESCRIPTION:
Glaucoma is the leading cause of irreversible blindness in China, as elsewhere in the world. In Chinese rural settings, where topical glaucoma medication is unlikely to be a practical and sustainable option, surgery is the primary treatment modality for glaucoma. However, it is known that vision is quite likely to decline in the short to medium term after glaucoma surgery, and there are concerns that dis-satisfaction resulting from such vision changes might lead to negative social marketing, affecting uptake not only of glaucoma surgical care but other eye operations (principally cataract) as well. We propose to test the impact on post-operative satisfaction of a multi-media educational intervention designed to give patients a realistic expectation of their post operative course: glaucoma surgery is being performed NOT to improve vision, but do protect it from future harm, and vision may in fact decline for several weeks post operatively. A randomized controlled design will be used, and subjects undergoing glaucoma surgery will be enrolled at 4 rural county hospitals in rural Guangdong province, and randomized to receive the intervention or usual care. The principal outcome will be subjective satisfaction on a previously-tested questionnaire instrument, administered pre-operatively and post-operatively on two occasions in the first month following surgery. Patients not returning post-operatively to the surgical facility will be contacted by telephone for administration of the questionnaire. Other facility- and patient-related clinical and personal factors expected to influence satisfaction will also be recorded, and adjusted for in all analyses.

ELIGIBILITY:
Inclusion Criteria:

* age≥18 years, glaucoma patients who do the peripheral iridectomy or trabeculotomy

Exclusion Criteria:

* patients who had been the trabeculotomy, vision≤0.05, severe psychotic disorders and dysgnosia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
The mean satisfaction score over three follow-up visits | 1 week, 2 week and 4 week after surgery.
  The primary outcome is the mean satisfaction score calculated by adding up the satisfaction scores at three follow-up visits: 1 week, 2 week and 4 week after surgery and dividing the total by the number of scores. The satisfaction score was assessed as a cumulative score.
  Composite outcome, in which multiple end points are combined, are frequently used as primary outcome measures in randomized trials and are often associated with increased statistical efficiency, although such measure may prove challenging for the interpretation of results. (Freemantle N, Calvert M, Wood J, Eastaugh J, Griffin C. Composite outcomes in randomized trials: greater precision but with greater uncertainty? JAMA. 2003; 289: 2554-2559)

SECONDARY OUTCOMES:
The rate of willingness to recommend surgery to a friend or relative with glaucoma | 1 week, 2 week and 4 week after surgery.
  The measurement method:questionnaire
Personality in both groups using Eysenck Personality Questionnaire-Revised Short Scale for Chinese (EPQ-RSC) access glaucoma patients personality | before surgery
Knowledge scores about glaucoma | before surgery and 1 week, 2 week and 4 week after surgery
Intraocular pressure in both groups | before surgery and 1 week, 2 week and 4 week after surgery
  Unit of Intraocular pressure is mmHg.
visual acuity in both groups | before surgery and 1 week, 2 week and 4 week after surgery
  Visual acuity testing use Snellen-based letter charts,such as a Snellen score of 6/12 (20/40), indicating an observer can resolve details as small 2 minutes of visual angle, corresponds to a LogMAR of 0.3 (since the base-10 logarithm of 2 is 0.3)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Congdon, MD,MPH, Principal Investigator — The Key Laboratory,Zhongshan Ophthalmic Center,Sun Yat-sen University
Locations (1):
- Blindness Preventment and Treatment Department, Guangzhou, Guangdong, China